CLINICAL TRIAL: NCT05849545
Title: Comparing the Effects of the Graston Tool and Neuromuscular Reeducation in Reducing Cervical Headache.
Brief Title: Effects of Garston Tool and Neuromuscular Reeducation in Cervical Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Jaweria Syed
Record Dates: First submitted 2022-12-23; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston Tool (Experimental): Graston instrument, 20 strokes per minute proximal to distal and 20 strokes per minute distal to proximal for a period of 3 minutes was given over the painful area. GT group protocol included the use application of IASTM along with the application of ice therapy at the end of the session. The assessment of patients was done at the initial and last visit before the completion of the treatment program. Three treatment sessions per week were given to each patient for a total of four weeks.
  Interventions: Device: Garston tool
- Neuromuscular Re-Education (Active Comparator): General stretching and strengthening exercises for the neck muscles. The protocol of treatment for the NMR group included the use of the Neuromuscular re-education soft tissue mobilization technique (NMR) followed by active movements of the patient.
  Interventions: Procedure: Neuromuscular Re-education

INTERVENTIONS:
Device: Garston tool — GT group protocol included the use application of IASTM along with the application of ice therapy at the end of the session. Using the Graston instrument, 20 strokes per minute proximal to distal and 20 strokes per minute distal to proximal for a period of 3 minutes were given over the painful area. Baseline values were recorded for demographics evaluation and episodes of pain onsets. The assessment of patients was done at the initial and last visit before the completion of the treatment program. Three treatment sessions per week were given to each patient for a total of four weeks.
  Other Names: Neuromuscular Re-education
  Arms: Graston Tool
Procedure: Neuromuscular Re-education — General stretching and strengthening exercises for the neck muscles. The protocol of treatment for the NMR group included the use of the Neuromuscular re-education soft tissue mobilization technique (NMR) followed by active movements of the patient.
  Arms: Neuromuscular Re-Education

SUMMARY:
Patients suffering from Cervicogenic headache have restricted range of motion and pain which in turn causes functional disability and reduced quality of life. The aim of this research was to determine the effects of Graston technique to improve range of motion, function, and reduction of pain and in patients having Cervicogenic headache

DETAILED DESCRIPTION:
A randomized controlled trial in which Graston Technique and Neuromuscular Re-education technique would be applied on patients presenting with cervicogenic headaches by using different tools and the changes would be examined pre and post intervention. The participants fulfilling inclusion criteria would be randomly allocated to two groups. Both groups received different protocols and will be assessed on data collection tool on their first and last visit using Goniometer, Headache Disability Index (HDI), Neck pain Disability Index (NDI) and Numeric Pain Rating Scale (NPRS). Participants of both groups will be pre-tested before the application of interventional techniques and post-tested after the application of respective intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: Minimum 20years- Maximum 50 years (Male/Female)
* Unilateral pain
* Neck stiffness and ROM restrictions
* Pain exacerbated by posture and neck movements
* Pain effecting QOL
* Positive flexion-rotation test

Exclusion Criteria:

* Headache not of cervical origin
* Congenital condition of cervical spine
* Headache with autonomic involvement, dizziness or visual impairment
* Inability to tolerate the flexion rotation test
* Conditions contraindicated for graston technique

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in pain on 10 points on Numeric Pain Rating Scale at 4th week | Baseline and 4th week
  The Numeric Pain Rating Scale, is a validated, self reported tool assessing average pain intensity over period of last 24 hours. Possible pain ranges from 0( No pain) to 10 (Worst pain).
  Change= (Week 4 Score - Baseline Score )
Change from Baseline in pain on 27 items on Headache Disability Index at 4th week | Baseline and 4th week
  Headache Disability Index is a 27 items questionnaire that identify the limitations experienced due to headache. It includes questions to identify the frequency ranges from one per month, more than one but less than four per months, more than one per week and intensity of headache ranges from mild to moderate and to severe.
Change from Baseline in pain on 10 items on Neck Disability Index at 4th week | Baseline and 4th week
  Neck Pain Disability Index is a 10 items questionnaire that identify the functional status of patients based on their conditions. it includes questions related to pain, personal care, reading, lifting, headaches, driving, sleeping , work, focus and leisure.

CONTACTS AND LOCATIONS:
Overall Officials: Nazma Namroz, Principal Investigator — Riphah International Univeristy, Islamabad
Locations (1):
- Nazma, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
there is a plan
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Elsocht G, Delaunaij T, Van Durme M, Van Hautegem E. Cervicogenic Headache.
- [Background] Biondi DM. Cervicogenic headache: a review of diagnostic and treatment strategies. J Am Osteopath Assoc. 2005 Apr;105(4 Suppl 2):16S-22S. PMID 15928349
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743
- [Background] Fredriksen TA, Antonaci F, Sjaastad O. Cervicogenic headache: too important to be left un-diagnosed. J Headache Pain. 2015;16:6. doi: 10.1186/1129-2377-16-6. Epub 2015 Jan 20. PMID 25604994
- [Background] Warren 1. Hammer M D, DABCO. Functional Soft-Tissue Examination and Treatment by Manual Methods 2007 2007.
- [Background] Portillo-Soto A, Eberman LE, Demchak TJ, Peebles C. Comparison of blood flow changes with soft tissue mobilization and massage therapy. J Altern Complement Med. 2014 Dec;20(12):932-6. doi: 10.1089/acm.2014.0160. PMID 25420037
- [Background] Stow R. Instrument-assisted soft tissue mobilization. International journal of athletic therapy and training. 2011;16(3):5-8.
- [Background] Hall TM, Robinson KW, Fujinawa O, Akasaka K, Pyne EA. Intertester reliability and diagnostic validity of the cervical flexion-rotation test. J Manipulative Physiol Ther. 2008 May;31(4):293-300. doi: 10.1016/j.jmpt.2008.03.012. PMID 18486750
- [Background] Sandmark H, Nisell R. Validity of five common manual neck pain provoking tests. Scand J Rehabil Med. 1995 Sep;27(3):131-6. PMID 8602474
- [Background] Page P. Cervicogenic headaches: an evidence-led approach to clinical management. Int J Sports Phys Ther. 2011 Sep;6(3):254-66. PMID 22034615
- [Background] Racicki S, Gerwin S, Diclaudio S, Reinmann S, Donaldson M. Conservative physical therapy management for the treatment of cervicogenic headache: a systematic review. J Man Manip Ther. 2013 May;21(2):113-24. doi: 10.1179/2042618612Y.0000000025. PMID 24421621
- [Background] Schoensee SK, Jensen G, Nicholson G, Gossman M, Katholi C. The effect of mobilization on cervical headaches. J Orthop Sports Phys Ther. 1995 Apr;21(4):184-96. doi: 10.2519/jospt.1995.21.4.184. PMID 7773270
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Boyer S, Novack J, Madsen L, Kingma J, Schrader J, Docherty C. The Immediate Effects of Graston Technique© on Hamstring Flexibility Compared to a Control. Journal of Athletic Training. 2017;52(6):S94.
- [Background] Barger KM. Compressive versus decompressive soft tissue therapy on acute hamstring flexibility and pain in male athletes with perceived hamstring tightness: Oklahoma State University; 2016.
- [Background] Cheatham SW, Lee M, Cain M, Baker R. The efficacy of instrument assisted soft tissue mobilization: a systematic review. J Can Chiropr Assoc. 2016 Sep;60(3):200-211. PMID 27713575